CLINICAL TRIAL: NCT06148402
Title: Fruquintinib Plus Camrelizumab and Capecitabine as Salvage Therapy After Progression on FOLFOXIRI-based First-line Treatment in Patients With Unresectable/Metastatic Colorectal Cancer: a Prospective Phase II Study
Brief Title: Fruquintinib Plus Camrelizumab and Capecitabine as Salvage Therapy After Progression on FOLFOXIRI-based First-line Treatment in Patients With Unresectable/Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2023-1049-01
Record Dates: First submitted 2023-11-03; First posted 2023-11-28 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Unresectable/Metastatic Colorectal Cancer
Keywords: Fruquintinib; Camrelizumab; Capecitabine; mCRC; salvage therapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013; camrelizumab; Capecitabine

STUDY DESIGN:
Intervention Model Description: fruquintinib 5 mg once daily, 2 weeks on/1 week off, plus camrelizumab 200 mg Q3W and capecitabine 750mg/square meter twice, 2 weeks on/1 week off, q3w
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fruquintinib plus camrelizumab and capecitabine (Experimental): fruquintinib 5 mg once daily, 2 weeks on/1 week off, plus camrelizumab 200 mg Q3W and capecitabine 750mg/square meter twice, 2 weeks on/1 week off, q3w
  Interventions: Drug: Fruquintinib plus camrelizumab and capecitabine

INTERVENTIONS:
Drug: Fruquintinib plus camrelizumab and capecitabine — fruquintinib 5 mg once daily, 2 weeks on/1 week off, plus camrelizumab 200 mg Q3W and capecitabine 750mg/square meter twice, 2 weeks on/1 week off, q3w

SUMMARY:
FOLFOXIRI-based regimen is more used as a first-line therapeutic approach for patients diagnosed with unresectable or metastatic colorectal cancer for its superior efficacy. However, there are no standard recommendations for second-line therapy after progression on FOLFOXIRI with or without targeted therapy. Here, the investigators conduct this open-label, single arm phase II study to evaluate whether fruquintinib in combination with camrelizumab and capecitabine can be the salvage therapy following FOLFOXIRI based regimen for mCRC. Patients diagnosed with unresectable or metastatic colorectal cancer progression on FOLFOXIRI-based regimen are included;or patients have progression or untolerated toxicity with irinotecan, oxaliplatin and fluorouracil successively within one year; patients with BRAF mutation were allowed to receive BRAF inhibitor therapy with or without MEK inhibitor therapy after FOLFOXIRI-based regimen.

Patients participated in this study will receive fruquintinib 5 mg once daily, 2 weeks on/1 week off, plus camrelizumab 200 mg Q3W and capecitabine 750mg/square meter twice, 2 weeks on/1 week off, repeated every three weeks. The primary endpoint is Objective Response Rate(ORR). The investigators estimated that 30 patients were necessary. Secondary endpoints include progression-free survival, overall survival, safety, and exploratory ctDNA for efficacy prediction for unresectable or metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic or locally advanced, unresectable colorectal cancer confirmed by histology or cytology
2. The occurrence of metastases after radical resection of colorectal cancer does not require additional histological or cytological confirmation unless more than 5 years since surgery for the primary tumor
3. Progression or toxicity intolerance of first-line treatment with or without targeted drugs (bevacizumab or cetuximab) with FOLFOXIRI regimen or the sequential administration of irinotecan, oxaliplatin, and fluorouracil within a year; if patients with BRAF mutations, who have been treated with BRAF inhibitor alone or in combination with MEK inhibitor also can be included.
4. Target lesion defined by the Response Evaluation Criteria in Solid Tumor (RECIST criteria)
5. Age ≥18 years old, performance status (ECOG) score ≤ 2
6. Estimated expectancy life at least 12 weeks
7. Adequate blood, liver and kidney function, as follows:

   1. Hemoglobin ≥8g/dl,
   2. neutrophil absolute count ≥1000/μL,
   3. platelets ≥ 75,000 /μL;
   4. Total bilirubin ≤1.5 x upper limit of normal (ULN),
   5. alkaline phosphatase, aspartate aminotransferase (AST (SGOT) and alanine aminotransferase (ALT (SGPT)) ≤2.5 x ULN (if liver metastasis is present, ≤5 x ULN),
   6. Serum creatinine ≤1.5 x ULN or calculated creatinine clearance >50mL/min (calculated according to Cockcroft Gault formula),
   7. urinary protein excretion (if protein >30 mg/dL or 2+, 24-hour urinary protein quantity must ≤1g)
8. International Normalized Ratio (INR) or activated partial thromboplastin time (APTT) <1.5 x ULN (thromboembolic event must be ruled out if D-dimer is abnormal)
9. Negative pregnancy test within 7 days before enrollment; Pregnancy tests can only be omitted in women who do not have any reproductive potential (e.g., postmenopausal women who had amenorrhea ≥2 years or prior hysterectomy or bilateral oophorectomy). Fertile wo-men and men must consent to the use of appropriate contraception at the time of enrollment and during study participation. If a woman becomes pregnant or suspects that she is pregnant while participating in this study, she must notify her physician immediately; Breastfeeding women must be excluded
10. Consent to provide blood samples for specific relevant analyses
11. Have the ability to understand and sign the written informed consent

Exclusion Criteria:

1. Received antitumor chemotherapy or biotherapy within 28 days prior to the first use of the investigational drug. The exception is a single dose of radiotherapy up to 8Gy for pain relief of non-target lesion during the first 14 days of enrollment
2. Untreated or symptomatic brain metastases
3. The exclusion criteria of fruquintinib are as follows:

   1. History of heart disease: Congestive heart failure (CHF) grade II or higher, according to the New York Heart Association (NYHA); Active coronary artery disease and myocardial infarction within 6 months prior to study initiation; New angina or unstable angina (occurrence at rest) that have not been evaluated within 3 months; arrhythmias that require antiarrhythmic therapy; except in participants who have been treated and who the investigator believes have stable/controlled disease;
   2. Uncontrolled hypertension (systolic blood pressure >150 mmHg or diastolic blood pressure >90 mmHg) and a history of hypertensive crisis or hypertensive encephalopathy;
   3. History of arterial thrombosis or embolism events (within 6 months)
   4. Critical vascular diseases (such as aortic aneurysm, aortic dissection, symptomatic peripheral vascular disease)
   5. People with bleeding tendency or coagulation disorder
   6. Had major surgery (including open biopsy, severe trauma, etc.) within 14 days prior to study enrollment, or expected to require major surgery during the study period, and had minor surgery (excluding Implantable Venous Access Port or peripherally inserted central venous catheter) within 7 days prior to study enrollment
   7. Abdominal fistula, gastrointestinal perforation, peptic ulcer or abdominal abscess in the past 6 months
   8. Severe, non-healing wounds, ulcers or fractures
   9. History of posterior reversible encephalopathy syndrome
   10. previous treatment with fruquintinib;
4. Inability to swallow tablets, malabsorption syndrome or any condition affecting gastrointestinal absorption; Patients with incomplete obstruction/obstruction syndrome/intestinal obstruction signs/symptoms at initial diagnosis may be admitted to the study if they have received definitive treatment (such as surgical) to resolve symptoms;
5. Active autoimmune disease or history of autoimmune disease with possible recurrence (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism [controllable only by hormone replacement therapy can be included]); Participants with non-systemic skin diseases such as vitiligo, psoriasis, and alopecia, type 1 diabetes controlled with insulin, or asthma in complete remission in childhood without any intervention as adults can be enrolled; Patients with asthma requiring medical intervention with bronchodilators are excluded;
6. Immunosuppressive or systemic hormone therapy for immunosuppressive purposes (dose >10mg/ day prednisone or other therapeutic hormone) within 14 days prior to initiation of study therapy
7. Severe infection within 4 weeks prior to initiation of study treatment, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia; Oral or intravenous administration of therapeutic antibiotics within 2 weeks prior to initiation of study treatment (patients receiving prophylactic antibiotics, for example, to prevent urinary tract infections or exacerbation of chronic obstructive pulmonary disease are eligible for study participation)
8. Patients with congenital or acquired immune deficiency (such as HIV infection)
9. Have received live attenuated vaccines within 28 days prior to initiation of study treatment, or are expected to require such vaccines during camrelizumab treatment or within 60 days after the last administration of camrelizumab
10. According to the investigator's judgment, the patient has other factors that may affect the study results or lead to the forced termination of the study, such as alcoholism, drug abuse, other serious diseases，including mental illness，requiring combined treatment, serious laboratory abnormalities, and family or social factors which will affect the safety of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Undergo imaging examination to evaluate efficacy every 6 weeks ±7 days, and every 9 weeks ±7 days in the second year (up to 2 years)
  Objective Response Rate is defined as the percentage of patients relative to the total of enrolled subjects who achieve a complete response (CR) or partial response (PR) based on CT or MRI scan images confirmed 4-6weeks later.

SECONDARY OUTCOMES:
Progression-free survival | Undergo imaging examination to evaluate efficacy every 6 weeks ±7 days, and every 9 weeks ±7 days in the second year (up to 2 years)
  Progression-free survival is defined as the time from study enrollment to first disease progression or death, whichever occurs first
Overall survival | from the date of enrollment to the date of death from any cause，assessed up to 2 years
  Overall survival is defined as the time from study enrollment to the date of death due to any cause
Adverse Events and Serious Adverse Events | from the date of the first medicine to 28days after the last medicine，assessed up to 2 years
  Assessment of Safety and tolerance for Fruquintinib plus camrelizumab and capecitabine as salvage therapy in patients with unresectable/metastatic colorectal cancer，including incidence, severity and outcomes of adverse events (AEs) and categorized by severity in accordance with the NCI CTCAE Version 5.0.
Circulating tumor DNA(ctDNA) and efficacy | from the date of enrollment to the date of progression，assessed up to 2 years
  Explore the correlation between dynamics of serum ctDNA and efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Qiong Yang, doctor, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guo Y, Zhang W, Ying J, Zhang Y, Pan Y, Qiu W, Fan Q, Xu Q, Ma Y, Wang G, Guo J, Su W, Fan S, Tan P, Wang Y, Luo Y, Zhou H, Li J. Phase 1b/2 trial of fruquintinib plus sintilimab in treating advanced solid tumours: The dose-escalation and metastatic colorectal cancer cohort in the dose-expansion phases. Eur J Cancer. 2023 Mar;181:26-37. doi: 10.1016/j.ejca.2022.12.004. Epub 2022 Dec 13. PMID 36628898
- [Background] Garcia-Alfonso P, Benavides M, Falco E, Munoz A, Gomez A, Sastre J, Rivera F, Montagut C, Salgado M, Lopez-Ladron A, Lopez R, Ruiz de Mena I, Duran G, Aranda E; Spanish Cooperative Group for the Treatment of Digestive Tumors (TTD). Single-Agent Regorafenib in Metastatic Colorectal Cancer Patients with Any RAS or BRAF Mutation Previously Treated with FOLFOXIRI plus Bevacizumab (PREVIUM Trial). Oncologist. 2018 Nov;23(11):1271-e128. doi: 10.1634/theoncologist.2018-0316. Epub 2018 Aug 17. PMID 30120161
- [Background] Rossini D, Lonardi S, Antoniotti C, Santini D, Tomasello G, Ermacora P, Germani MM, Bergamo F, Ricci V, Caponnetto S, Moretto R, Zaniboni A, Pietrantonio F, Buonadonna A, Ritorto G, Masi G, Latiano TP, Rapisardi S, Falcone A, Cremolini C. Treatments after progression to first-line FOLFOXIRI and bevacizumab in metastatic colorectal cancer: a pooled analysis of TRIBE and TRIBE2 studies by GONO. Br J Cancer. 2021 Jan;124(1):183-190. doi: 10.1038/s41416-020-01089-9. Epub 2020 Oct 7. PMID 33024268
- [Background] Loupakis F, Cremolini C, Masi G, Lonardi S, Zagonel V, Salvatore L, Cortesi E, Tomasello G, Ronzoni M, Spadi R, Zaniboni A, Tonini G, Buonadonna A, Amoroso D, Chiara S, Carlomagno C, Boni C, Allegrini G, Boni L, Falcone A. Initial therapy with FOLFOXIRI and bevacizumab for metastatic colorectal cancer. N Engl J Med. 2014 Oct 23;371(17):1609-18. doi: 10.1056/NEJMoa1403108. PMID 25337750
- [Background] Mettu NB, Ou FS, Zemla TJ, Halfdanarson TR, Lenz HJ, Breakstone RA, Boland PM, Crysler OV, Wu C, Nixon AB, Bolch E, Niedzwiecki D, Elsing A, Hurwitz HI, Fakih MG, Bekaii-Saab T. Assessment of Capecitabine and Bevacizumab With or Without Atezolizumab for the Treatment of Refractory Metastatic Colorectal Cancer: A Randomized Clinical Trial. JAMA Netw Open. 2022 Feb 1;5(2):e2149040. doi: 10.1001/jamanetworkopen.2021.49040. PMID 35179586